CLINICAL TRIAL: NCT01538875
Title: Hydralazine vs. Labetalol for the Management of Hypertensive Crisis in Patients With Hypertensive Disorders of Pregnancy. A Randomized Controlled Trial.
Brief Title: Hydralazine Versus Labetalol for the Management of Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research and Development, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2012-06
Record Dates: First submitted 2012-02-18; First posted 2012-02-24 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension, Pregnancy Induced
Keywords: Hypertension, pregnancy induced; Hydralazine; Labetalol
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Hydralazine; Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydralazine (Experimental): Patients with an hypertensive crisis during pregnancy will receive 5mg IV every 15 minutes (Maximum number of doses: 3).
  Interventions: Drug: Hydralazine
- Labetalol (Active Comparator): Patients with an hypertensive crisis during pregnancy will receive 20 mg of Labetalol IV. After 15 minutes if the crisis continue, 40 mg IV. After 15 minutes if the crisis continue, 80 mg IV. Then, if the crisis continue, 80 mg IV every 15 minutes (maximum dose: 300 mg IV in total).
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Hydralazine — Patients with an hypertensive crisis during pregnancy will receive 5mg IV every 15 minutes until high blood pressure is controlled (Maximum number of doses: 3).
  Arms: Hydralazine
Drug: Labetalol — Patients with an hypertensive crisis during pregnancy will receive 20 mg of Labetalol IV. After 15 minutes if the crisis continue, 40 mg IV. After 15 minutes if the crisis continue, 80 mg IV. Then, if the crisis continue, 80 mg IV every 15 minutes (maximum dose: 300 mg IV in total).
  Arms: Labetalol

SUMMARY:
Hypertensive crisis (defined as a systolic pressure > 160mmHg or a diastolic pressure > 110mmHg) in patients with a hypertensive disorder of pregnancy is a serious complication with severe and even deadly consequences. The management in this population had been studied, but no consensus has been reached with regards to which treatment is better. Our study will compare two drugs: Hydralazine and Labetalol for the management of hypertensive crisis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 24 weeks.
* Hypertensive Crisis (systolic pressure > 160 mmHg / diastolic pressure < 110mmHg).

Exclusion Criteria:

* Known allergy to hydralazine.
* Known allergy to labetalol.
* Severe Bradycardia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Control of Hypertensive Crisis | 10 months
  Number of patients with hypertensive crisis in which the blood pressure is controlled with the use of the assigned drug, without requiring additional medications.

SECONDARY OUTCOMES:
Adverse reactions | 10 months
  Number of patients in each group that reported an adverse reaction to the drug assigned.
Number of doses | 10 months
  Number of doses of the assigned drug required to lower blood pressure, without requiring additional medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama